CLINICAL TRIAL: NCT04863469
Title: Neurocognitive Optimization and Enhancement for Brain Health and Performance
Brief Title: Brain-Physical Optimization Conditioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2751
Record Dates: First submitted 2020-11-12; First posted 2021-04-28 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Physical Performance
Keywords: cognitive fatigue; demand; endurance performance; perceived exertion; effort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-POC high load Intervention (Experimental): aerobic exercise [heartrate range (HRR) 70-75% of max HR, on treadmill] and a computerized high-load task for 45 minutes, 3 times per week, for 6 weeks
  Interventions: Behavioral: B-POC high load intervention
- B-POC low load intervention (Sham Comparator): aerobic exercise [heartrate range (HRR) 70-75% of max HR, on treadmill] and a computerized low-load task for 45 minutes, 3 times per week, for 6 weeks
  Interventions: Behavioral: B-POC low load intervention

INTERVENTIONS:
Behavioral: B-POC high load intervention — aerobic exercise [heartrate range (HRR) 70-75% of max HR, on treadmill] and a computerized high-load task for 45 minutes, 3 times per week, for 6 weeks
  Arms: B-POC high load Intervention
Behavioral: B-POC low load intervention — aerobic exercise [heartrate range (HRR) 70-75% of max HR, on treadmill] and a computerized low-load task for 45 minutes, 3 times per week, for 6 weeks
  Arms: B-POC low load intervention

SUMMARY:
Brain-Physical Optimization Conditioning (B-POC) aims to enhance physical performance by expanding the traditional focus of endurance training from purely physical training to the domain of cognitive endurance (Staiano et al., 2015; Dallaway et al., 2017). The current study seeks to isolate neurocognitive mechanisms of performance, particularly under high stress (e.g., physical or cognitive load) conditions, and to develop corresponding cognitive optimization tools.

DETAILED DESCRIPTION:
Brain-Physical Optimization Conditioning (B-POC) aims to enhance physical performance by expanding the traditional focus of endurance training from purely physical training to the domain of cognitive endurance (Staiano et al., 2015; Dallaway et al., 2017). B-POC uses an acute mentally fatiguing task during routine exercise with the aim of optimizing the effects of physical endurance (e.g., aerobic exercise). B-POC differs from other types of cognitive training by increasing the cognitive demands of a specific concurrent task rather than teaching a cognitive strategy and relying on task transfer effects. Similar to strengthening a muscle, cognitive trainings may be one means of increasing Soldier's cognitive capacity and improving performance (Walton et al., 2018).

ELIGIBILITY:
Inclusion Criteria:

* Healthy active duty Soldiers
* 18-40 years old
* Available for study duration

Exclusion Criteria:

* Failure of an Army Physical Fitness/Combat Test (APFT/ACFT) test
* On a physical profile that prevents them from 1) engaging in intense aerobic exercise, 2) running on a treadmill, 3) riding the stationary bike, and 4) performing a cognitive task on a computer screen.
* Medically non-deployable
* Impaired cognitive function due to medication, injury or illness,
* Have been advised by a medical professional not to engage in aerobic exercise
* Are a pregnant female

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Time to Failure Test | 7 weeks
  The Time to Failure Test (TFT) requires participants to run on a treadmill with increases in either grade (0.5% increase) and speed (~0.3-0.5 mph) every two minutes in an alternating format for the first 16 minutes, after which settings remain constant until self termination of the exercise. The TFT settings (work rate) are calculated from an individual's last 2 mile run time. Physiological load (heart rate, oxygen consumption) and perceived exertion (RPE) are measured throughout the TFT.
  The primary outcome is change in time to failure (minutes, seconds) on the endurance test from baseline to post0test (~7 weeks).

SECONDARY OUTCOMES:
Dynamic Marksmanship | Pre-to-post ruck time (~30-90 minutes)
  The Dynamic Marksmanship Test requires participants to complete four increasingly difficult phases of target identification (friend vs. foe) and elimination using a rifle marksmanship simulator (EST). The test is completed both before and after a 3-mile ruck march, which is completed with +30% bodyweight. Physiological output (HR), and subjective ratings of workload (NASA-TLX) are assessed throughout each marksmanship test.
  The primary outcome is change in accuracy (%) from pre-ruck performance to post-ruck performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Directorate - West, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No